CLINICAL TRIAL: NCT04330807
Title: Physiopathology of Neuromuscular Function Related to Fatigue in Chronic Renal Disease
Acronym: PIONEER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Collaborators: Le Mans Universite (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHM-2020/S8/01
Record Dates: First submitted 2020-03-26; First posted 2020-04-02 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Stage 3B; Chronic Kidney Disease stage4; Chronic Kidney Disease Stage 5; Fatigue
Keywords: Neuromuscular abilities; Dynapenia; Over-60-year-old patients
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fatigue | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with chronic kidney disease (Other): Patients will perform a Handgrip fatigability test with their dominant hand and will complete two questionnaires of assessment of subjective fatigue.
  Interventions: Other: Handgrip fatigability test; Other: Questionnaires
- CONTROL GROUP (Other): Patients will perform a Handgrip fatigability test with their dominant hand and will complete two questionnaires of assessment of subjective fatigue.
  Interventions: Other: Handgrip fatigability test; Other: Questionnaires

INTERVENTIONS:
Other: Handgrip fatigability test — Dynamometric and electromyographic assessment: patient is sitting on a chair, back upright, humerus vertically placed and forearm landing parallel to a support. Dominant arm is chosen for test and electrodes placement.
  The assessment is divided in 4 phases for a total of 30 minutes duration: Warm-up, determination of reference force settings (fast sub-maximal contractions and maximal voluntary contractions), fatigability period and rest.
Other: Questionnaires — Assessment of subjective fatigue with Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) and Multidimensional Fatigue Inventory (MFI-20) questionnaires

SUMMARY:
Chronic Kidney Disease (CKD) induces many metabolic troubles especially for the advanced CKD (stage 3b-5) patients and their prevalence and importance grow with the deterioration of the glomerular filtration rate (GFR). Among them, muscle wasting is common and multifactorial, partially explained by an imbalance between protein catabolism and synthesis. Muscular strength is also affected beyond the reduction of the lean body mass, resulting in profound fatigue.

The present study seeks to quantify the prevalence of low muscular strength production (dynapenia) in a cohort of elderly patients with advanced CKD, through a maximal voluntary contraction (MVC) handgrip test compared to control data available in the literature, matched in term of age and sex. It also aims to investigate the link between the reported fatigue (subjective) and the evolution of the MVC, called critical force (fcrit) during a fatiguing task (objective fatigability).

ELIGIBILITY:
Inclusion Criteria:

* Adults, aged 60 and over
* Social security coverage
* Signed informed consent
* For patient with Chronic Kidney Disease, estimated glomerular filtration rate (eGFR) less than 45ml/min/1.73m2 (Stage 3b) for at least 3 months
* For patient with Chronic Kidney Disease, stable clinical condition (i.e., Creatinine increased by a maximum of 25% in the previous 3 months)
* For control group, 1:1 recruitment with case matching with CDK patients on gender (i.e., male and female) and the presence of diabètes (i.e., presence and absence)
* For control group, blood test with control of renal function available and dated less than 6 months: with eGFR > 60ml/min/1.73m2 (and control of glucose or glycated hemoglobin for diabetic controls)

Exclusion Criteria:

* Pregnant women
* Under guardianship or minor
* Neuromuscular disease
* Dementia
* Upper limbs history of surgery or pathologies preventing from fitting EMG electrodes or measuring handgrip force
* Life expectancy of less than 3 months estimated by medical judgment
* Programed hospitalization in the previous 3 months
* Participation to another interventional clinical trial
* Acute kidney disease
* On dialysis or expected start of dialysis within next 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
DYNAPENIA | 1 day
  The main outcome of the study is to defined the prevalence of dynapenia for advanced CKD elderly patients. Dynapenia will be established when the mean of the first three MVC of the protocol is lower compared to the reference values appaired for age and sex. For reference values of elderly, please see Ramírez-Vélez et al., (2019).

SECONDARY OUTCOMES:
EMG signal | 1 day
  To analyze the amplitude of the EMG signal recorded, it will be rectified with the Root Mean Square (RMS) method. Frequency analysis will be performed with the Fast Fourier Transform (FFT).
Objective fatigue | 1 day
  The nmF is an indicator of the objective fatigue, it is identified by measuring the Fcrit during the fatigability period of the protocol (Figure 1). The value of Fcrit is the asymptote of the MVC curve plotted. This value is calculated for each individual.
Subjective fatigue | 1 day
  The symptom of fatigue will be assessed with two questionnaires, the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) and the Multidimensional Fatigue Inventory (MFI-20). FACIT-F is a validated questionnaire in French language (Kwakkenbos et al., 2014), slightly short, including 13 pragmatically and simple affirmations (e.g., I am too tired to eat) with Likert scale (0: "Not at all" to 4: "enormously"). The questionnaire depicted 4 dimensions (i.e., General fatigue, mental fatigue, reduced activities, motivation) and the final score ranges from 0 to 52, with an elevated score depicted a low fatigue. MFI-20 is a validated questionnaire in French language (Gentile et al., 2003) focused about fatigue. It is built with a balance between positive trend questions (e.g., Physically I feel I am in an excellent condition) and negative trend question (e.g., Physically I feel only able to do a little). An elevated score depicted a higher fatigue.

OTHER OUTCOMES:
Anthropometric data | Within 3 months for the CKD patients, within 6 months for the control volunteers.
  Only relevant data will be collected from medical folder such as age, sex... to determine anthropometric data.
Clinical data | Within 3 months for the CKD patients, within 6 months for the control volunteers.
  Relevant data will be collected from medical folder such as existence of a diabetes, type of kidney disease, time of follow-up, Charlson Comorbidity Index (CCI ; Charlson et al., 1987) and Malnutrition Inflammation Score (Borges et al., 2017) to determine comorbidities data.
Nutritional data | Within 3 months for the CKD patients, within 6 months for the control volunteers.
  Relevant data will be collected from medical folder such as Malnutrition Inflammation Score (Borges et al., 2017), Subjective global assessment, albumin, total cholesterol, HDL, LDL, triglycerides, uric acid, blood formula count, creatinine, urea, glycemia, 24 hours proteinuria, pre-albumine, uric acid to determine nutritional status.
Biochemical data | Within 3 months for the CKD patients, within 6 months for the control volunteers.
  Relevant data will be collected from medical folder such as calcium, phosphorus, PTH, vitamin D, bicarbonate, sodium and potassium to define biochemical data.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chatrenet A, Beaune B, Fois A, Pouliquen C, Audebrand JM, Torreggiani M, Paris D, Durand S, Piccoli GB. PhysIOpathology of NEuromuscular function rElated to fatigue in chronic Renal disease in the elderly (PIONEER): study protocol. BMC Nephrol. 2020 Jul 25;21(1):305. doi: 10.1186/s12882-020-01976-6. PMID 32711479